CLINICAL TRIAL: NCT03298295
Title: A Pilot Study for the Systematic Evaluation of the Inflammatory Response to Commercially Available Insulin Infusion Catheters in Subcutaneous Adipose Tissue
Brief Title: Inflammatory Response to CSII Catheters in a Tummy Tuck Model
Acronym: IRCATT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRCATT
Record Dates: First submitted 2017-09-21; First posted 2017-10-02 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus; Insulin Pump Therapy; Continuous Subcutaneous Insulin Infusion
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Non-diabetic patients scheduled for selective plastic surgery (abdominoplasty).
Masking Description: The only person blinded in this study is the pathologist analyzing the tissue sections.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Insertion of Insulin Infusion Catheters (Experimental): Non-diabetic patients scheduled for abdominoplasty will be inserted continuous subcutaneous insulin infusion (CSII) catheters of two different materials into the part of the abdomen which will be removed during surgery.
  Interventions: Device: Continous Subcutaneous Insulin Infusion Catheter

INTERVENTIONS:
Device: Continous Subcutaneous Insulin Infusion Catheter — Catheters will be inserted into the abdomen of each patient using aseptic technique according to the following schedule: (1) 8 days before surgery, (2) 4 days before surgery and (3) 1 day before surgery (Table 1). At each time point 2 steel (Medtronic Sure-T, 9 mm) and 2 Teflon (Medtronic Quick-set®, 9 mm) CSII catheters will be inserted into the subcutaneous abdominal tissue. In total, 12 catheters will be inserted into each patient's abdomen using only the area predefined by the plastic surgeon for removal.

SUMMARY:
In insulin pump therapy, insulin is continuously infused into the subcutaneous adipose tissue via a continuous subcutaneous insulin infusion (CSII) catheter using a basal/bolus pattern. Unfortunately, insulin absorption from the tissue surrounding a CSII catheter can be slow, variable, and unreliable. It is recommended to replace CSII catheters after 2 to 3 days of use. Frequently changing the injection site can be tedious and moreover leads to scarring, while reusing the same injection site can lead to medical complications such as lipohypertrophy. CSII catheters are manufactured from both steel and Teflon and use of either of these materials is based on personal preference/experience rather than scientific, empirical data. We hypothesize that the inflammatory response to CSII catheters is a major contributor to variable insulin absorption and that this response is significantly different between materials and catheters shapes. In order to develop CSII catheters with an extended life-time up to 7 days, we need to better understand the inflammatory response caused by the introduction and maintenance of a CSII catheter into the subcutaneous adipose tissue. This study is a pilot study in humans scheduled for elective plastic surgery where a large skin flap is removed from the abdominal region. Teflon and steel CSII catheters will be inserted into the abdomen 7, 4, and 3 days prior to surgery. This study design allows for the removal of tissue plugs surrounding CSII catheters without causing additional scarring for the patient.

DETAILED DESCRIPTION:
Background:

Approximately one million patients worldwide manage their diabetes with an insulin pump. Insulin is continuously infused into the subcutaneous adipose tissue via a Continuous Subcutaneous Insulin Infusion (CSII) catheter using a basal/bolus pattern that can be adjusted by the patient according to meal times, mimicking the natural function of the pancreas. One major advantage of this form of therapy is the improvement of living quality. Compared to multiple daily insulin injections, the catheter has to be inserted only once every 2-3 days where it remains within the subcutaneous tissue. This is especially advantageous for children of young age.

Unfortunately, insulin absorption from the tissue surrounding a CSII catheter can be slow, variable, and unreliable. It is recommended to replace infusion sets and CSII catheters after 2 to 3 days of clinical use. After this time, blood glucose control becomes difficult for the patient because insulin absorption from the subcutaneous tissue into the blood stream and lymphatics becomes highly variable.

The underlying mechanisms for impaired insulin absorption are poorly understood and the knowledge of rotating the site of injection is based on user experience. Frequently changing the injection site can be tedious and moreover leads to scarring, while reusing the same injection site can lead to medical complications such as lipohypertrophy. In order to develop CSII catheters with an extended life-time up to 7 days, there is a need to better understand the inflammatory response caused by the introduction and maintenance of a CSII catheter into the subcutaneous adipose tissue. The clinical use of a 7-day CSII catheter with low pharmacokinetics (PK) variability will significantly improve blood glucose control, decrease the risk for hypoglycemia, increase compliance, and decrease cost. Since continuous glucose monitoring (CGM) devices are approved for 7-day wear time, the development of a CSII catheter with extended lifetime is also crucial for the development of single-port artificial pancreas (AP) systems where CSII and CGM are combined in one catheter, mimicking pancreatic function. Furthermore, the improvement of catheter longevity will reduce insertion sites and scars. This is especially important for children with a smaller body surface area.

The choice of one material over the other is largely based on the patient's personal preference, his or her endocrinologist's or diabetes educator's opinion and therapy costs. There is a trend in both the United States and Europe towards using Teflon sets (90 % and 75 %, respectively) but approximately 40 to 45 % of pump users in Germany use steel catheters. Compared to Teflon, steel catheters are easier to insert and are less prone to kinking, and can be worn by patients allergic to Teflon. Patients using steel catheters report better metabolic control, less variable insulin absorption and less unexplained hyperglycemia (Heinemann 2016; Reichert et al. 2013). However, especially during exercise, steel may cause discomfort and the softer and more flexible Teflon catheter is assumed to be more comfortable to wear. The wear-time of the CSII catheter considerably varies between patients (from 2 to 10 days), although recommendations for the optimal frequency of changing an insulin infusion set (2 days for steel and 3 days for Teflon) exist.

In a prior pig study the inflammatory response to commercial CSII catheters comparing steel, Teflon and Teflon with an anti-inflammatory coating was analyzed. There was significant reduction in area of inflammation and macrophage recruitment around the non-coated and coated Teflon catheters. Steel elicited the most severe inflammatory response with significantly higher fibrosis.

Although the pig has proven to be an excellent model for the study of human skin and adipose tissue, there is an urgent medical need to confirm these findings in a human model. For the histopathological and molecular analysis of subcutaneous tissue in the vicinity of the catheter, large amounts of tissue need to be excised from the site of interest. This makes a human study almost impossible. Nevertheless, the generation of human data is crucial and a lot of this important information is still lacking in diabetes research and treatment. The possibility to excise extensive amounts of tissue without causing additional scars or pain (except that caused by the abdominoplasty itself) for the patient presents the main benefit of this study setup.

Aim:

The aim of this study is to compare the inflammatory response to commercially available CSII catheters of two different materials (steel and Teflon) over 1 day, 4 days and 7 days of wear-time in humans scheduled for elective plastic surgery (abdominoplasty).

Hypothesis:

Conventional steel CSII catheters elicit a more severe acute inflammatory response in the subcutaneous adipose tissue than Teflon CSII catheters.

H0 = there is no difference in mean area of fibrin deposition around catheters H1 = there is a significant difference in mean area of fibrin deposition between catheters

ELIGIBILITY:
Inclusion Criteria:

* Men and women, age 18 years or older
* Scheduled elective abdominoplasty at the Dpt. of Plastic Surgery, Medical University of Graz
* Signed informed consent form

Exclusion Criteria:

* Allergy to Teflon or steel
* Known skin diseases (atopic dermatitis, psoriasis)
* History of immunodeficiency diseases
* Patients on glucocorticoid or other immunomodulating therapy
* History of bleeding disorder
* Pregnancy or planned pregnancy
* Unable to fully understand study procedures and to provide informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Area of inflammation (mm2) | 7 days
  Assessed by microscopy; area of inflamed tissue, including cell infiltration, necrosis, fibrin/collagen deposition

SECONDARY OUTCOMES:
Area of fibrin deposition (mm2) | 7 days
  Assessed by microscopy; area of fibrin
Area of fat necrosis (mm2) | 7 days
  assessed by microscopy; area of necrosed adipocytes
Inflammation distance (mm) | 7 days
  assessed by microscopy; distance from skin surface to lowest point of microscopically assessed inflammation
Cytokine gene expression (fold change) | 7 days
  Assessed by qPCR; relative fold change in gene expression compared to non-traumatized tissue (IL-1b, TNFa, TGFb, IL-6, IL-8, IL-10)
Macrophage marker gene expression (fold change) | 7 days
  Assessed by qPCR; relative fold change in CD68 gene expression compared to non-traumatized tissue

CONTACTS AND LOCATIONS:
Overall Officials: Lars-Peter Kamolz, MD Prof, Principal Investigator — Medical University of Graz
Locations (1):
- Division of Plastic, Aesthetic and Reconstructive Surgery, Graz, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Conwell LS, Pope E, Artiles AM, Mohanta A, Daneman A, Daneman D. Dermatological complications of continuous subcutaneous insulin infusion in children and adolescents. J Pediatr. 2008 May;152(5):622-8. doi: 10.1016/j.jpeds.2007.10.006. Epub 2008 Jan 22. PMID 18410763
- [Background] Deiss D, Adolfsson P, Alkemade-van Zomeren M, Bolli GB, Charpentier G, Cobelli C, Danne T, Girelli A, Mueller H, Verderese CA, Renard E. Insulin Infusion Set Use: European Perspectives and Recommendations. Diabetes Technol Ther. 2016 Sep;18(9):517-24. doi: 10.1089/dia.2016.07281.sf. Epub 2016 Aug 15. PMID 27526329
- [Background] Facchinetti A, Sparacino G, Guerra S, Luijf YM, DeVries JH, Mader JK, Ellmerer M, Benesch C, Heinemann L, Bruttomesso D, Avogaro A, Cobelli C; AP@home Consortium. Real-time improvement of continuous glucose monitoring accuracy: the smart sensor concept. Diabetes Care. 2013 Apr;36(4):793-800. doi: 10.2337/dc12-0736. Epub 2012 Nov 19. PMID 23172973
- [Background] Heinemann L. Insulin Infusion Sets: A Critical Reappraisal. Diabetes Technol Ther. 2016 May;18(5):327-33. doi: 10.1089/dia.2016.0013. Epub 2016 Feb 17. PMID 26885764
- [Background] Heinemann L, Fleming GA, Petrie JR, Holl RW, Bergenstal RM, Peters AL. Insulin pump risks and benefits: a clinical appraisal of pump safety standards, adverse event reporting, and research needs: a joint statement of the European Association for the Study of Diabetes and the American Diabetes Association Diabetes Technology Working Group. Diabetes Care. 2015 Apr;38(4):716-22. doi: 10.2337/dc15-0168. PMID 25776138
- [Background] Heinemann L. Variability of insulin absorption and insulin action. Diabetes Technol Ther. 2002;4(5):673-82. doi: 10.1089/152091502320798312. PMID 12450450
- [Background] Heinemann L, Krinelke L. Insulin infusion set: the Achilles heel of continuous subcutaneous insulin infusion. J Diabetes Sci Technol. 2012 Jul 1;6(4):954-64. doi: 10.1177/193229681200600429. PMID 22920824
- [Background] Heinemann L, Walsh J, Roberts R. We Need More Research and Better Designs for Insulin Infusion Sets. J Diabetes Sci Technol. 2014 Mar;8(2):199-202. doi: 10.1177/1932296814523882. Epub 2014 Feb 27. No abstract available. PMID 24876567
- [Background] Macmillan K, Bruera E, Kuehn N, Selmser P, Macmillan A. A prospective comparison study between a butterfly needle and a Teflon cannula for subcutaneous narcotic administration. J Pain Symptom Manage. 1994 Feb;9(2):82-4. doi: 10.1016/0885-3924(94)90160-0. PMID 8021539
- [Background] Pickup JC, Yemane N, Brackenridge A, Pender S. Nonmetabolic complications of continuous subcutaneous insulin infusion: a patient survey. Diabetes Technol Ther. 2014 Mar;16(3):145-9. doi: 10.1089/dia.2013.0192. Epub 2013 Nov 1. PMID 24180294
- [Background] Reichert, D. et al., 2013. Realität der Insulinpumpentherapie in Diabetesschwerpunktpraxen: Daten von 1142 Patienten aus 40 diabetologischen Schwerpunktpraxen. Diabetes Stoffwechsel Herz, 22, pp.367-375.
- [Background] Sampson Perrin AJ, Guzzetta RC, Miller KM, Foster NC, Lee A, Lee JM, Block JM, Beck RW; T1D Exchange Clinic Network. A web-based study of the relationship of duration of insulin pump infusion set use and fasting blood glucose level in adults with type 1 diabetes. Diabetes Technol Ther. 2015 May;17(5):307-10. doi: 10.1089/dia.2014.0336. Epub 2015 Jan 26. PMID 25622214
- [Background] Schmid V, Hohberg C, Borchert M, Forst T, Pfutzner A. Pilot study for assessment of optimal frequency for changing catheters in insulin pump therapy-trouble starts on day 3. J Diabetes Sci Technol. 2010 Jul 1;4(4):976-82. doi: 10.1177/193229681000400429. PMID 20663464
- [Background] Sullivan TP, Eaglstein WH, Davis SC, Mertz P. The pig as a model for human wound healing. Wound Repair Regen. 2001 Mar-Apr;9(2):66-76. doi: 10.1046/j.1524-475x.2001.00066.x. PMID 11350644
- [Background] Walsh J, Roberts R, Weber D, Faber-Heinemann G, Heinemann L. Insulin Pump and CGM Usage in the United States and Germany: Results of a Real-World Survey With 985 Subjects. J Diabetes Sci Technol. 2015 Jun 12;9(5):1103-10. doi: 10.1177/1932296815588945. PMID 26071425